CLINICAL TRIAL: NCT05652075
Title: Efficacy and Safety of Ultrasound Guided Combined Pericapsular Nerve Group Block and Lateral Femoral Cutaneous Nerve Versus Lumbar Plexus Block for Postoperative Analgesia After Total Hip Arthroplasty: Randomized Clinical Study.
Brief Title: PENG and LFCN Block Versus Lumbar Plexus Block for Postoperative Analgesia After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 473:10/2022
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain; Regional Block
Keywords: PENG; lumber plexus; hip surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG and LFCN (Experimental)
  Interventions: Procedure: pericapsular nerve group and lateral femoral cutaneous nerve block
- lumbar plexus (Experimental)
  Interventions: Procedure: lumbar plexus block

INTERVENTIONS:
Procedure: pericapsular nerve group and lateral femoral cutaneous nerve block — Will undergo pericapsular nerve group block (PENG) combined with lateral femoral cutaneous nerve under ultrasound guided block with 20 mL of 0.25% bupivacaine.
  Arms: PENG and LFCN
Procedure: lumbar plexus block — Will undergo Lumbar plexus block (LPB) under ultrasound guided block with 20 mL of 0.25 % bupivacaine.
  Arms: lumbar plexus

SUMMARY:
Regional anesthesia for postoperative analgesia in THA includes epidural anesthesia and peripheral nerve blocks. However epidural anesthesia has a great role in THA, it has become restricted as perioperative antithrombotic drugs are generally used for orthopedic patients.

the study aim to evaluate and compare efficacy and safety of pericapsular nerve group block (PENG) block and lateral femoral cutaneous nerve versus Lumbar plexus block on postoperative analgesia in hip surgery.

ELIGIBILITY:
Inclusion Criteria:

(ASA) physical status I to III scheduled for hip surgery aged (30-70) years

Exclusion Criteria:

* Drug allergy,
* Morbid obesity (BMI >40 kg/m2),
* Coagulopathy,
* Psychiatric disorder,
* Opioid dependence,
* Patient refusal to give informed consent.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale pain scores | 24 hour
  pain score from 0-10 which 0 mean no pain and 10 the worst pain

SECONDARY OUTCOMES:
first analgesic request | 24 hour
  time to demand nalbuphine
total analgesic consumption | 24 hour
  total nalbuphine in mg consumed in the first day
First time to ambulate | 24 hours
  first time to move

CONTACTS AND LOCATIONS:
Overall Officials: hassan m. hetta, lecturer, Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No